CLINICAL TRIAL: NCT02587754
Title: Acupuncture in the Treatment of Fatigue in Parkinson's Disease: a Pilot Randomized Controlled Study
Brief Title: Acupuncture in the Treatment of Fatigue in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-10-16; First posted 2015-10-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease; Fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: 2 arm study comparing acupuncture with sham
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum acupuncture (Active Comparator): 10 sessions of verum acupuncture
  Interventions: Device: Acupuncture
- Placebo acupuncture (Placebo Comparator): 10 sessions of placebo acupuncture via use of placebo acupuncture needles
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — 10 sessions of acupuncture, twice a week over 5 weeks.

SUMMARY:
This study evaluates the efficacy of acupuncture in the treatment of fatigue in participants with Parkinson's Disease. Half of participants will receive real acupuncture while the half will receive placebo acupuncture.

DETAILED DESCRIPTION:
This will be a single centre, single blinded 2-group randomized controlled study, with participants receiving either verum acupuncture or placebo acupuncture.

A retractable non-invasive placebo needle will be used in the placebo arm. Both the real and placebo needles have a fine needle body and copy handle and look exactly the same. However, the placebo needle has a retractable shaft and blunt tip. When pressed onto the skin, it telescopes into the handle and the blunt tip stays on the skin instead of penetrating it. The plastic tube with adhesive foot-plate is placed on the skin to hold it in place. The real needle, on the other hand, has a normal sharp tip which allows it to pierce the skin.

The following acupoints will be needled: Stomach 36 (bilateral), Spleen 6 (bilateral), Kidney 3 (bilateral), Large Intestine 4 (bilateral), Pericardium 6 (bilateral), and Conception Vessel 6. These points were chosen based on Traditional Chinese Medicine theory (which attributed fatigue to deficiencies of spleen, kidney and qi).

Each acupuncture session will be based on a strict protocol, and conversation between acupuncturists and participants will be kept to a minimum.

Participants will be assessed at 3 intervals:

1. Week 0 (baseline)
2. Week 5 (completion of intervention)
3. Week 9 (4 weeks after completion of intervention

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD based on criteria developed by Gelb et al which is adopted by the National Institute of Neurological Disorders and Stroke, US National Institute of Health.
2. Age 21-85 years old
3. Presence of persistent fatigue of a moderate level for at least 4 weeks' duration. Moderate fatigue is defined as a score of ≥10 on the general fatigue domain of the Multidimensional Fatigue Inventory.
4. No acupuncture treatment in the past 6 months.

Exclusion Criteria:

1. Significant cognitive, language or psychiatric illnesses which prevents the subject from understanding instructions and participating in the study.
2. Needle phobia
3. Comorbidity with a bleeding disorder
4. Known anemia with hemoglobin level less than 10g/dl.
5. Known congestive cardiac failure and/or end stage renal disease
6. Female subjects of childbearing age
7. Presence of symptomatic postural hypotension

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
General Fatigue score of the Multidimensional Fatigue Inventory | General Fatigue score of the Multidimensional Fatigue Inventory at week 5
  Measure of fatigue

SECONDARY OUTCOMES:
General Fatigue score of the Multidimensional Fatigue Inventory | General Fatigue score of the Multidimensional Fatigue Inventory at week 9
  Measure of fatigue
Unified Parkinson's Disease Rating Scale (UPDRS) | UPDRS score at week 5
  Measure of severity of Parkinson's Disease
Unified Parkinson's Disease Rating Scale (UPDRS) | UPDRS score at week 9
  Measure of severity of Parkinson's Disease
Parkinson's Disease Questionnaire-39 (PD 39). | PD 39 score at week 5
  Measure of quality of life
Parkinson's Disease Questionnaire-39 (PD 39). | PD 39 score at week 9
  Measure of quality of life
Geriatric Depression Scale (GDS) | GDS score at week 5
  Measure of depression
Geriatric Depression Scale (GDS) | GDS score at week 9
  Measure of depression

OTHER OUTCOMES:
Adverse events | Adverse events will be captured up to 9 weeks
  all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Keng H Kong, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore